CLINICAL TRIAL: NCT05867095
Title: Targeted Abdominal Lymph nodE Dissections Randomized for Surgical NavigaTion (TALENT)
Brief Title: Navigated Abdominal Lymph Node Dissections
Acronym: N16LND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N16LND
Record Dates: First submitted 2022-11-09; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Image-guide Surgery; Lymph Node Metastasis
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Surgery, Computer-Assisted; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation (Experimental): Patients will get the standard of care in the Netherlands with the addition of surgical navigation
  Interventions: Procedure: Surgical navigation
- Conventional (Other): Patients will get the standard of care in the Netherlands
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: Surgical navigation — Patients will be operated with assistance of a navigation system
  Arms: Navigation
Procedure: Conventional — Patients will be operated using the conventional technique
  Arms: Conventional

SUMMARY:
Image-guided navigation surgery allows for full utilization of pre-operative imaging during surgery, and has the potential of reducing both irradical resections and morbidity. In this study we will randomize patients which will undergo an abdominal lymph node dissection in order to evaluate the actual technical and clinical benefit of navigation

DETAILED DESCRIPTION:
In the study patients will be randomized between the use of a surgical navigation system or not. The operation itself will be performed according to current clinical practice, and the navigation system will be used for better localization and orientation during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for open abdominal surgery in which targeted removal of one or more pathological lymph nodes is part of the surgical plan

Exclusion Criteria:

* Metal implants in the pelvic area
* Contra-indication for contrast enhanced CT scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Number of failed procedures | 3 months
  Failed procedure is defined as: presence of any residual target lymph node on follow-up imaging

SECONDARY OUTCOMES:
Surgical time to remove lymph node | After surgery
  time from having the surgical field prepared for lymph node localization to actual removal of the lymph node, overall surgical time,
LN success | 3 months
  individual LN retrieval rate

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groen HC, Wit EMK, Heerink WJ, Kuhlmann KFD, Nijkamp JA, van Veen R, Schoots IG, Balduzzi S, Zijlmans HJMAA, van Leeuwen PJ, van der Poel HG, Ruers TJM. Surgical navigation for targeted retroperitoneal lymph-node removal: a randomised, controlled, phase 3 trial. EClinicalMedicine. 2024 Jul 26;74:102754. doi: 10.1016/j.eclinm.2024.102754. eCollection 2024 Aug. PMID 39737148